CLINICAL TRIAL: NCT04081025
Title: A 10 Year Longitudinal Study of Oral Health and Risk Factors for Oral Disease
Brief Title: Oral Health and Risk Factors for Oral Disease
Status: Completed | Type: Observational
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Kristina Edman, Principal Investigator, Dalarna County Council, Sweden
Other Study IDs: EpiWux
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Periodontal Diseases; Dental Caries; Quality of Life
MeSH Terms: conditions — Periodontal Diseases; Dental Caries | interventions — Oral Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Age Groups 35, 50, 65, 75 and 85
  Interventions: Other: EpiWux

INTERVENTIONS:
Other: EpiWux — A cross-sectional and longitudinal study including a questionnaire and a clinical examination
  Other Names: Oral Health

SUMMARY:
Oral health has improved considerably in recent decades in Sweden, as well as in other countries. However, despite great improvements with regard to periodontal disease and dental caries in recent decades, global problems still persist, and as a consequence of retaining natural teeth high up in age, the risk for oral disease increases.

DETAILED DESCRIPTION:
Traditionally, the number of teeth has been a measure of good oral health, and the World Health Organization (WHO) stipulated goals of a minimum of 20 functional teeth at the age of 80 years have been reached in some industrialized countries. Oral Health means more than good teeth and is integral to general health. The relationship between oral and general health has been recognized. For example, periodontal disease is associated with diabetes and rheumatoid arthritis. The severity of periodontal disease and number of teeth have been associated with an increased burden of cardiovascular disease.

There is a lack of longitudinal studies of oral Health and risk factors for oral disease.

ELIGIBILITY:
Inclusion Criteria:

* None

Exclusion Criteria:

* None

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals in age Groups 35, 50, 65, 75 and 85 years
Sampling Method: Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Periodontal disease | 10 years (2008-2018)
  The severity of alveolar bone loss are based on bone levels at interproximal sites as seen on radiographs in the premolar and molar regions in both jaws. The diagnostic categories are (1)'no bone loss', defined as normal alveolar bone height in the molar and premolar regions (i.e., a distance ≤2 mm between the cemento-enamel junction and the alveolar bone crest (2) moderate bone loss, defined as alveolar bone loss >2 mm but not exceeding one-third of the length of the roots, or if angular bony defects/furcation defects degree II and III are present on two to three teeth in the molar-premolar region; and (3)'severe bone loss', defined as alveolar bone loss exceeding one-third of the length of the roots, or if angular bony defects/furcation defects degree II and III are present on more than three teeth in the molar and premolar regions.
Periodontal disease | At one occasion (2018)
  The severity of alveolar bone loss are based on bone levels at interproximal sites as seen on radiographs in the premolar and molar regions in both jaws. The diagnostic categories are (1)'no bone loss', defined as normal alveolar bone height in the molar and premolar regions (i.e., a distance ≤2 mm between the cemento-enamel junction and the alveolar bone crest (2) moderate bone loss, defined as alveolar bone loss >2 mm but not exceeding one-third of the length of the roots, or if angular bony defects/furcation defects degree II and III are present on two to three teeth in the molar-premolar region; and (3)'severe bone loss', defined as alveolar bone loss exceeding one-third of the length of the roots, or if angular bony defects/furcation defects degree II and III are present on more than three teeth in the molar and premolar regions.
Risk factors for periodontal disease | Ten years (2008-2018)
  A questionnaire is used to assess risk factors for periodontal disease.The outcome variables is: Education:
  * Up to secondary school
  * University or college of higher learning
  Economy for dental care:
  * No limited financial resources for dental care
  * Limited financial resources for dental care
  Marital status:
  * Married/cohabitant
  * Single living
  Tobacco use:
  * Current smoker
  * Former smoker
Dental caries | 10 years (2008-2018)
  Number of teeth with dental caries
Dental caries | At one occasion (2018)
  Number of teeth with dental caries
Risk factors for dental caries | Ten years (2008-2018)
  Number of teeth with dental caries
Oral Health Related Quality of Life | One occasion (2018)
  A 9-item survey instrument (Oral Impact on Daily Performance), using a five-point Likert scale, ranging from "never" (1), "less than once a month (2), 1-2 times a month (3), 1-2 times a week (4), and "every, or nearly every day" (5) was used.
  The questions are as follows: "during the past 6 months, how often have problems with your mouth or teeth caused any difficulty with:
  * Eating and enjoying food
  * Speaking
  * Pronouncing clearly
  * Doing light physical activities
  * Cleaning teeth
  * Sleeping and relaxing
  * Smiling, laughing and showing teeth without embarrassment
  * Maintaining usual emotional state without being irritable
  * Carrying out major work or social role and enjoying contact with people

CONTACTS AND LOCATIONS:
Overall Officials: Karin Gunnars Hellgren, Study Chair — Region Dalarna
Locations (1):
- Kristina Edman, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided